CLINICAL TRIAL: NCT06905158
Title: Evaluating the Effectiveness of a Non-invasive Tinnitus Device in Reducing Symptoms of Tinnitus and Mental Health Difficulties in Military Veterans: A Pilot Randomised Controlled Trial
Brief Title: Evaluation of a Non-invasive Tinnitus Device for the Management of Tinnitus Symptoms in Military Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Combat Stress (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No ID yet
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Tinnitus
Keywords: Tinnitus; Non-invasive device; Sound therapy; Tinnitus device; White noise device; Military veterans
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Waitlist-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate intervention arm (Experimental): All participants will receive the non-invasive device to their registered address and will be asked to use it for a period of one month. This will involve wearing the device around ones neck or body during the day and docking it at night for 24/7 relief. Participants can alter the volume and frequency of the device to fit into their individual experience.
  Interventions: Device: White noise device
- Waitlist control arm (Other): The WL control group will receive the device one-month post-randomisation
  Interventions: Device: White noise device

INTERVENTIONS:
Device: White noise device — * Product name: TinniSoothe white noise-non-invasive tinnitus device
  * Usage: Worn around the neck during the daytime and docked to a stand at night
  * Duration: At least one-month of use
  Other Names: TinniSoothe; Non-invasive white noise device; Tinnitus sound device

SUMMARY:
The prevalence of tinnitus in military veterans is notably higher than the non-veteran population and can significantly disrupt the lives of veterans. Given the profound impact of tinnitus on the lives of veterans, along with the considerable economic burden and barriers to treatment, it is crucial to explore the feasibility of new approaches. Wearable sound technologies offer a non-invasive and easily accessible approach. As such, this waitlist-controlled trial aims to assess the efficacy of this new non-invasive white noise wearable device in reducing tinnitus symptoms between baseline and the one-month post-randomisation among veterans who have experienced tinnitus for at least three months.

DETAILED DESCRIPTION:
The presence of tinnitus has been significantly associated with depression, anxiety, sleep difficulties and job performance in addition to poorer general physical health.. However, to our knowledge, there is currently no intervention for tinnitus that is supported as effective for most people. As such, there is a need to explore alternative approaches. Sound therapy offers an easily accessible, non-invasive, low-cost option. As such, this study aims to explore the effectiveness of a non-invasive white noise device in reducing symptoms of tinnitus and mental health difficulties in military veterans. A total of 20 military veterans who have self-reported experiencing tinnitus for at least three months will be recruited. : In this waitlist-controlled trial, the tinnitus device will be compared to the waitlist-controlled group who will receive the device one-month post-randomisation. The trial will be conducted in a veteran population (n = 20) that was recruited from a prior study that had aimed to explore the impact of tinnitus on wellbeing within a veteran population. Once the participants receive the tinnitus device, they will be asked to use the device for a period of one month. The primary outcome is the change in self-reported tinnitus symptoms and mental health difficulties between baseline (day 0) and the one-month post-randomisation (day 28). The outcome variables of interest will be assessed at all timepoints (baseline, one-month post-randomisation, and two-months post-randomisation) and the predictor variables will only be assessed at baseline to reduce participant burden. It is hypothesised that the non-invasive device will result in significant reductions in symptoms of tinnitus (as indicated using the TFI) and mental health difficulties (as measured using the gHQ-12) from baseline to one-month post-intervention in comparison to a waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in speaking and reading English.
* United Kingdom Armed Forces veteran
* Persistent tinnitus for at least three months (participants with tinnitus had to confirm experience of constant ringing or buzzing [bilateral or unilateral] lasting longer than three months).
* Able to receive the TinniSoothe device to their registered address
* Able to follow study instructions
* Sign the written consent form prior to any study-related procedures being performed

Exclusion Criteria:

* Below 18 years of age
* Significant severe hearing loss without hearing aids
* Individuals who have already habituated to tinnitus
* Veterans receiving concurrent treatment for tinnitus (e.g., other wearable devices or ongoing audiological therapies)
* Active self-harm or suicidal ideation
* Severe psychotic disorder, dissociative identity disorder or other severe mental health difficulty
* Current alcohol or drug-use disorder or dependency requiring further support or treatment that would significantly impact treatment engagement, as assessed clinician
* Unwilling and/or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms of tinnitus measured using the Tinnitus Functional Index (TF) | [Time Frame: Change from baseline TFI score at one-month post-randomisation and two-months post-randomisation]
  Scores range from 0-250, with higher scores indicating greater tinnitus symptoms
Symptoms of mental health difficulties measured using the General Health Questionnaire-12 | [Time Frame: Change from baseline General Health Questionnaire-12 score at one-month post-randomisation and two-months post-randomisation]
  Scores range from 0-36, with higher scores indicating greater psychological distress

SECONDARY OUTCOMES:
Satisfaction of life as measured using the Satisfaction with life Scale (SWLS) | [Time Frame: Change from baseline SWLS score at one-month post-randomisation and two-months post-randomisation]
  Scores range from 5-35, with a higher score indicating greater life satisfaction.
Sleep as measured using the Insomnia Severity Index (ISI) | [Time Frame: Change from baseline ISI score at one-month post-randomisation and two-months post-randomisation]
  Scores range from 0-28, with a higher score indicating greater insomnia severity.

OTHER OUTCOMES:
Symptoms of PTSD as measured using the Posttraumatic Stress Disorder Checklist For Diagnostic and Statistical Manual of Mental Disorders-5- Short Version (PCL- 5-4) | [Time Frame: Predictor variable]
  A 4-item measure of the presence of PTSD symptoms according to the Diagnostic and Statistical Manual of Mental Disorders-IV. Scores range from 0-16, with a higher score indicating more severe PTSD
Physical health and somatic symptoms as measured using the Patient Health Questionnaire-15 | [Time Frame: Predictor variable]
  Scores range from 0-30, with higher scores indicating greater severity of physical health and somatic symptoms
Qualitative questionnaire | [Time Frame: Consenting participants will be contacted at one-month post-randomisation for the immediate intervention group and two-months post-randomisation for the waitlist control group]
  Consenting participants will be contacted at one-month post-randomisation for the immediate intervention group and two-months post-randomisation for the waitlist control group
Retention rate | [Time Frame: Intervention end (approximately 1 year)]
  Feasibility endpoint
• Recruitment of target sample size (n = 20) | [Time Frame: Study end (approximately 1 year)]
  Feasibility endpoint
Incidence of adverse events across the duration of the study | [Time Frame: Study end (approximately 1 year)]
  Safety endpoint, calculated as total number of adverse events reported across the study. Adverse events as defined in the study protocol. Adverse events will be reported in the qualitative questionnaire post-intervention.

IPD SHARING:
Plan to Share IPD: No
No identifiable information will be shared with other researchers.